CLINICAL TRIAL: NCT02351973
Title: Comparison of Single and Combination Diuretics in Low-Renin Hypertension
Acronym: PATHWAY3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cambridge (Other)
Collaborators: University of Leicester (Other); University of Dundee (Other); University of Glasgow (Other); University of Edinburgh (Other); Imperial College London (Other); Barts & The London NHS Trust (Other); King's College London (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Morris Brown, Professor, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKCRN 4501; 2009-010068-41 (EudraCT Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amiloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hydrochlorthiazide (Active Comparator): Hydrochlorothiazide (HCTZ) ATC class: C03AA03 Form: Tablet Dose range: Phase 1: 25mg (2 x 12.5mg tablet) Phase 2: 50mg (4 x 12.5mg tablet) Maximum allowed dose: 50mg Administration: oral
  Interventions: Drug: Hydrochlorthiazide
- Amiloride (Active Comparator): Amiloride ATC class: C03DB01 Form: Tablet Dose range: Phase 1: 10mg (2 x 5mg tablet) Phase 2: 20mg (4 x 5mg tablet) Maximum allowed dose: 20mg Administration: oral
  Interventions: Drug: Amiloride
- Hydrochlorthiazide and Amiloride (Active Comparator): Hydrochlorothiazide (HCTZ) + Amiloride Form: Tablets (separate tablet of each drug) Dose range: Phase 1: HCTZ 12.5mg (1 tablet) + Amiloride 5mg (1 tablet) Phase 2: HCTZ 25mg (2 x 12.5mg tablet) + Amiloride 10mg (2 x 5mg tablet) Maximum allowed dose: HCTZ 25mg/ Amiloride 10mg Administration: oral
  Interventions: Drug: Hydrochlorthiazide and Amiloride

INTERVENTIONS:
Drug: Hydrochlorthiazide — HCTZ 25mg to 50mg All drugs will be provided in an acceptable container where the active agent is not identified on the drug label.
  In Phase 1 (weeks 0-12) patients will have 1 tablet from each of 2 bottles. These will contain either a) HCTZ 12.5mg in both bottles; b) amiloride 5mg in both bottles; OR c) one bottle of each.
  In Phase 2 (weeks13-24) patients will take 2 tablets from each of 2 bottles. These bottles will have the same contents as in Phase 1, except that the number of tablets will be twice as many.
  Arms: Hydrochlorthiazide
Drug: Amiloride — Amiloride 10mg to 20mg All drugs will be provided in an acceptable container where the active agent is not identified on the drug label.
  In Phase 1 (weeks 0-12) patients will have 1 tablet from each of 2 bottles. These will contain either a) HCTZ 12.5mg in both bottles; b) amiloride 5mg in both bottles; OR c) one bottle of each.
  In Phase 2 (weeks13-24) patients will take 2 tablets from each of 2 bottles. These bottles will have the same contents as in Phase 1, except that the number of tablets will be twice as many.
  Arms: Amiloride
Drug: Hydrochlorthiazide and Amiloride — HCTZ 12.5 to 25mg & + Amiloride 5mg to 10mg All drugs will be provided in an acceptable container where the active agent is not identified on the drug label.
  In Phase 1 (weeks 0-12) patients will have 1 tablet from each of 2 bottles. These will contain either a) HCTZ 12.5mg in both bottles; b) amiloride 5mg in both bottles; OR c) one bottle of each.
  In Phase 2 (weeks13-24) patients will take 2 tablets from each of 2 bottles. These bottles will have the same contents as in Phase 1, except that the number of tablets will be twice as many.
  Arms: Hydrochlorthiazide and Amiloride

SUMMARY:
The purpose of this study is to determine whether the routine combination of optimal thiazide and K+-sparing diuretic will both increase efficacy of BP reduction and reduce risk of glucose intolerance; and whether K+-sparing diuretics alone may have a neutral or even beneficial effect upon glucose tolerance.

DETAILED DESCRIPTION:
A major attraction of K+-sparing diuretics may be the absence of risk of new-onset diabetes (DM). Since they have not been compared in hypertension outcome trials, and DM has not been an endpoint in heart failure studies of spironolactone or eplerenone, we do not know for certain whether they are clean in this respect. Short-term studies suggest they are.49 Interestingly in INSIGHT there was no excess of DM in patients receiving HCTZ 25mg, which was combined with amiloride 2.5mg, but increased by 30% in patients on HCTZ/amiloride 50/5mg.44 In the proposed study we shall use the oral glucose tolerance test (OGTT) to provide an endpoint for each subject. This strategy has recently been employed to demonstrate a difference after just 12 weeks of dosing with a thiazide diuretic50. Hyperkalaemia has been the traditional concern about K+-sparing diuretics. We expect to demonstrate that in patients with eGFR ≥45, the risk of hyperkalaemia is nullified by combination with a thiazide. Instead then of amiloride being used mainly in trace doses to balance the hypokalaemia of thiazides, practice might reverse to thinking of thaizides as the "partner" used to negate risk of hyperkalaemia.

The challenge to designing this study is to compare several options among the diuretics while achieving clear cut answers to:

1. the comparison of combination with single diuretics and
2. the comparison of K+-sparing diuretics with thiazide.

A study of sufficient duration to establish efficacy and tolerability (especially upon glucose tolerance) cannot be crossover in design and therefore requires a large number of subjects to compare the options. In order to maximize recruitment whilst also maximizing sensitivity to detect changes in OGTT, we will open the trial to most of those patients with hypertension in whom diuretic is a reasonable next option, providing they have one feature of the metabolic syndrome - additional to hypertension.

ELIGIBILITY:
Inclusion Criteria;

Patients can proceed to placebo run-in if biochemical data available from previous 6 months, but cannot proceed to randomised treatment if eligibility not confirmed by baseline sample:

1. Age 18-80
2. Diagnosis of hypertension according to BHS criteria
3. Systolic BP on permitted background treatment ≥ 140 mmHg and home BP ≥ 130mmHg. Patients may be included if the PI anticipates BP criteria for inclusion will be met at randomisation
4. Indication for diuretic treatment:

   * Untreated + (age>55 AND/OR Black AND/OR renin<12mU/L)
   * receiving one or any permutation of the following: *ACEi, ARB, β-blocker, CCB, direct renin inhibitor
5. At least one other component (i.e. additional to hypertension) of the metabolic syndrome (reduced HDL, raised triglycerides, glucose, waist circumference)* * Definition of Metabolic Syndrome according to the International Diabetes Federation, 2006: Central obesity (waist circumference > 94cm male (>90 if Asian), > 80 female plus two of:

   * SBP ≥ 130 or DBP ≥ 85 mmHg
   * Fasting glucose >5.6mmol/l
   * Fasting Triglycerides > 1.7 mmol/l (or on rx)
   * HDL < 1.03 mmol/l males, < 1.29 mmol/l females (or on rx)

Exclusion Criteria:

1. Diabetes (types 1 or 2)
2. Secondary hypertension
3. eGFR < 45 mls/min
4. Plasma K+ outside normal range on two successive measurements during screening
5. Clinic SBP >200 mmHg or DBP >120mmHg, with PI discretion to override if home BP's lower
6. Requirement for diuretic therapy (other than for hypertension)
7. Absolute contra-indications to any of the study drugs
8. Current therapy for cancer
9. Anticipation of change in medical status planned surgical intervention requiring >2 weeks convalescence, actual or planned pregnancy)
10. Inability to give informed consent
11. Not on stable doses of all hypertensive medications to be continued throughout the study for a minimum of 4 weeks prior to randomisation, or not normally less than 2 weeks if early randomisation is required at the discretion of the PI.
12. Participation in a clinical study involving an investigational drug/device within 4 weeks of screening.
13. Any concomitant condition that may adversely affect the safety and/or efficacy of the study drug or severely limit the subject's lifespan or ability to complete the study
14. Treatment with any of the following prohibited medications:

    * Oral corticosteroids within 3 months of Screening and prohibited during study participation.
    * Chronic stable or unstable use of non-steroidal anti-inflammatory drugs other than acetylsalicylic acid is prohibited. Chronic use is defined as >3 consecutive or nonconsecutive days of treatment per week. intermittent use of NSAIDs is strongly discouraged throughout the duration of this study. If intermittent treatment is required, NSAIDs must not be used for more than a total of 2 days. For all subjects requiring analgesic or anti-pyretic agents, the use of paracetamol is recommended during study participation.
    * The use of short-acting oral nitrates (eg, sublingual nitroglycerin) is permitted; however, subjects should not take short-acting oral nitrates within 4 hours of Screening or any subsequent study visit.
    * The use of long-acting oral nitrates is permitted; however, the dose must be stable for at least 2 weeks prior to screening/ randomisation.
    * Use of sympathomimetic decongestants is permitted; but, not within 1 week prior to screening or randomisation. or within 1 day prior to study visits;
    * The use of theophylline is permitted; however, the dose must be stable for at least 4 weeks prior to Screening and throughout study participation.
    * The use of phosphodiesterase (PDE) type V inhibitors is permitted; however, subjects must refrain from taking these medications within 1 day of Screening or any subsequent study visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2009-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Blood glucose measured two hours after oral ingestion of a 75 G glucose drink, following overnight fasting. | 0, 12 and 24
  There will be hierarchical co-primary endpoints. First, the primary outcome (2hr glucose) will be compared between the amiloride and HCTZ cohorts. If amiloride is superior, a second primary analysis will compare cohorts on combination therapy and HCTZ. The analyses will adjust for baseline covariates.
  The difference in blood glucose, over the 6 months between baseline and the end of the study period, measured two hours after oral ingestion of a 75 g glucose drink, will be analysed using a mixed model with patients as a random effect. The model will include terms for gender, age, height, weight and smoking history.

SECONDARY OUTCOMES:
Home systolic BP. The secondary outcome is the difference from the end of placebo run-in to 24 weeks | 0, 12 and 24 weeks
Plasma insulin during OGTT. The secondary outcome is the change from end of placebo to 24 weeks in the rise in insulin from 0 to 30 minutes during oral glucose tolerance test | 0, 12 and 24 weeks
HbA1C. The secondary outcome is the change in HbA1c between end of placebo and 24 weeks | 0, 12, 24 weeks
Clinic systolic BP. The secondary outcome is the change in clinic systolic BP from end of placebo run-in to 24 weeks. | 0, 12, 24 weeks
Area under the curve of the oGTT. The secondary outcome is the difference in area under the curve of blood glucose, from 0-120 minutes after glucose ingestion, between the final day of the placebo run-in, and 24 weeks. | 0, 12, 24 weeks
Fasting serum lipids. The secondary outcome is the difference in fasting serum lipids, between the final day of the placebo run-in, and 24 weeks. | 0, 12, 24 weeks
The natriuretic response, as assessed from the compensatory increase in plasma renin. The secondary outcome is the difference in plasma renin from end of placebo run-in to 24 weeks | 0, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Professor MJ Brown, Principal Investigator — Cambridge University and Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Clinical Pharmacology Unit, Box 110, Level 3 ACCI, Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] NICE/BHS. CG34 Hypertension - NICE guideline (all the recommendations). http://www.nice.org.uk/guidance/CG34/niceguidance /pdf/english 2006
- [Background] Dickerson JE, Hingorani AD, Ashby MJ, Palmer CR, Brown MJ. Optimisation of antihypertensive treatment by crossover rotation of four major classes. Lancet. 1999 Jun 12;353(9169):2008-13. doi: 10.1016/s0140-6736(98)07614-4. PMID 10376615
- [Background] Deary AJ, Schumann AL, Murfet H, Haydock SF, Foo RS, Brown MJ. Double-blind, placebo-controlled crossover comparison of five classes of antihypertensive drugs. J Hypertens. 2002 Apr;20(4):771-7. doi: 10.1097/00004872-200204000-00037. PMID 11910315
- [Background] Taler SJ, Textor SC, Augustine JE. Resistant hypertension: comparing hemodynamic management to specialist care. Hypertension. 2002 May;39(5):982-8. doi: 10.1161/01.hyp.0000016176.16042.2f. PMID 12019280
- [Background] Kaplan NM. Resistant hypertension. J Hypertens. 2005 Aug;23(8):1441-4. doi: 10.1097/01.hjh.0000174968.72212.ac. PMID 16003165
- [Background] Black HR, Keck M, Meredith P, Bullen K, Quinn S, Koren A. Controlled-release doxazosin as combination therapy in hypertension: the GATES study. J Clin Hypertens (Greenwich). 2006 Mar;8(3):159-66; quiz 167-8. doi: 10.1111/j.1524-6175.2006.04811.x. PMID 16522992
- [Background] Law MR, Wald NJ, Morris JK, Jordan RE. Value of low dose combination treatment with blood pressure lowering drugs: analysis of 354 randomised trials. BMJ. 2003 Jun 28;326(7404):1427. doi: 10.1136/bmj.326.7404.1427. PMID 12829555
- [Background] Brown MJ, Cruickshank JK, Dominiczak AF, MacGregor GA, Poulter NR, Russell GI, Thom S, Williams B; Executive Committee, British Hypertension Society. Better blood pressure control: how to combine drugs. J Hum Hypertens. 2003 Feb;17(2):81-6. doi: 10.1038/sj.jhh.1001511. PMID 12574784
- [Background] Brown MJ, Palmer CR, Castaigne A, de Leeuw PW, Mancia G, Rosenthal T, Ruilope LM. Morbidity and mortality in patients randomised to double-blind treatment with a long-acting calcium-channel blocker or diuretic in the International Nifedipine GITS study: Intervention as a Goal in Hypertension Treatment (INSIGHT). Lancet. 2000 Jul 29;356(9227):366-72. doi: 10.1016/S0140-6736(00)02527-7. PMID 10972368
- [Background] Ramsay LE, Yeo WW, Jackson PR. Diabetes, impaired glucose tolerance and insulin resistance with diuretics. Eur Heart J. 1992 Dec;13 Suppl G:68-71. doi: 10.1093/eurheartj/13.suppl_g.68. PMID 1486909
- [Background] Bakris G, Molitch M, Hewkin A, Kipnes M, Sarafidis P, Fakouhi K, Bacher P, Sowers J; STAR Investigators. Differences in glucose tolerance between fixed-dose antihypertensive drug combinations in people with metabolic syndrome. Diabetes Care. 2006 Dec;29(12):2592-7. doi: 10.2337/dc06-1373. PMID 17130190
- [Derived] Brown MJ, Williams B, MacDonald TM, Caulfield M, Cruickshank JK, McInnes G, Sever P, Webb DJ, Salsbury J, Morant S, Ford I. Comparison of single and combination diuretics on glucose tolerance (PATHWAY-3): protocol for a randomised double-blind trial in patients with essential hypertension. BMJ Open. 2015 Aug 7;5(8):e008086. doi: 10.1136/bmjopen-2015-008086. PMID 26253567